CLINICAL TRIAL: NCT07224971
Title: Assessing the Impact of Circadian Rhythm on Anti-PD-1/PD-L1 Immunotherapy
Brief Title: Impact of Circadian Rhythm on Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liza Villaruz, MD (Other)
Responsible Party: Sponsor-Investigator, Liza Villaruz, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 25-127
Record Dates: First submitted 2025-10-31; First posted 2025-11-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced/Metastatic NSCLC
Keywords: anti-PD-1/PD-L1 Immunotherapy; Circadian Rhythm
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Immunotherapy dosing (Experimental): NSCLC and solid tumor patients who receive first-line or ICI therapy early in the day (prior to 11AM) versus late in the day (after 12PM) and NSCLC patients with stable or response disease after induction therapy receiving maintenance ICI therapy early in the day (prior to 11AM) versus late in the day (after 12PM)
  Interventions: Drug: Immunotherapy - PD-1 Blocker
- Late Immunotherapy dosing (Active Comparator): NSCLC and solid tumor patients who receive first-line or ICI therapy late in the day (started after 12 PM) and NSCLC patients with stable or response disease after induction therapy receiving maintenance ICI therapy late in the day (started after 12PM)
  Interventions: Drug: Immunotherapy - PD-1 Blocker

INTERVENTIONS:
Drug: Immunotherapy - PD-1 Blocker — Standard of Care Drugs (at investigator's discretion) may include: pembrolizumab, nivolumab, cemiplimab, durvalumab, dostarlimab, avelumab, and atezolizumab, or other immune checkpoint inhibitors used in cancer treatment that targets cancer cells by blocking the PD-1 receptor on T cells.

SUMMARY:
This study aims to determine whether morning versus afternoon treatment impacts efficacy of (standard of care) immunotherapy in a broad patient population. Patients with any type of advanced/metastatic malignancy are eligible to enroll in this study, as long as first-line anti-PD-1/PD-L1 immunotherapy is on label for their condition. Participants will then be randomized to either the early treatment group (administration must start and conclude by 11:00 AM +1 hour window) or the late treatment group (administration must start after 12:00 PM).

DETAILED DESCRIPTION:
The US market has many FDA approved options for anti-PD-1/PD-L1 immunotherapies, including pembrolizumab, nivolumab, cemiplimab, durvalumab, dostarlimab, avelumab, and atezolizumab, among others that are in development. With an estimated 56.55% of cancer patients eligible for treatment with anti-PD-1/PD-L1 immunotherapy (as of 2023), the impact of timing on immunotherapy efficacy should be delineated in order to provide the best care possible to patients This study will be implemented at a large regional cancer center in the United States. Three patient cohorts will be investigated: Non-Small Cell Lung Cancer (NSCLC) patients who receive first-line ICI therapy (Cohort A), NSCLC patients with stable disease or response after induction therapy receiving maintenance ICI therapy (Cohort B), and solid tumor patients receiving first-line ICI therapy (Cohort C).

To the best the knowledge of this principal investigator, this is the first prospective time-of-day immunotherapy study to take place in the US. Key endpoints include real-world progression free survival (rwPFS)[26], overall survival (OS), safety, quality of life (QoL), and pharmacoeconomic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort Specific Criteria

   * Cohort A: Advanced/metastatic NSCLC patients for which 1st line PD-1/PD-L1 therapy is on-label either alone or in combination.
   * Cohort B: Advanced/metastatic NSCLC patients who have completed up to 4 cycles of induction therapy who have stable disease or responsive disease and for which maintenance anti-PD-1/PD-L1 therapy is on-label either alone or in combination.
   * Cohort C: Advanced/metastatic solid tumor malignancy for which first-line anti-PD-1/PD-L1 therapy is on-label either alone or in combination.
2. Prior and concurrent therapy criteria

   o Patients should be ICI-naïve (this should be first-line therapy) (Cohorts A and C), or should have received ICI induction therapy and are now eligible for ICI maintenance therapy (Cohort B).
3. Must be willing to be randomized to complete therapy at assigned time of day, which may be early in the morning OR later in the day/into the evening.
4. Must be eligible to receive anti-PD-1/PD-L1 therapy singly or in combination with other FDA-approved agents according to standard of care practices, as determined by the clinical judgment of the investigator but according to approved label indications
5. Must have the ability to understand and the willingness to sign a written informed consent document.
6. Able to read and write in English.

Exclusion Criteria:

1. Participant unable to receive anti-PD-1/PD-L1 therapy due to prior allergic reactions to therapy or any therapy ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Real-world progression-free survival (rwPFS) - Cohort A | Up to 4.5 years
  Time from first dose of 1st line treatment to clinician documented clinical disease progression, initiation of new line of therapy, or death from any cause, whichever comes first. Real-world progression-free survival (rwPFS), defined as the time from first dose of 1st line treatment to clinician documented clinical disease progression, initiation of new line of therapy, or death from any cause, whichever came first. Per RECISIT v1.1, Progressive Disease: ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

SECONDARY OUTCOMES:
Overall Survival (OS) - Cohort A | Up to 4.5 years
  Overall Survival (OS) defined as time from first dose of 1st line treatment to death from any cause.
Real-world progression-free survival (rwPFS) - Cohort B | Up to 4.5 years
  Time from first dose of 1st line treatment to clinician documented clinical disease progression, initiation of new line of therapy, or death from any cause, whichever came first. Per RECISIT v1.1, Progressive Disease: ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Real-world progression-free survival (rwPFS) - Cohort C | Up to 4.5 years
  Time from first dose of 1st line treatment to clinician documented clinical disease progression, initiation of new line of therapy, or death from any cause, whichever came first. Per RECISIT v1.1, Progressive Disease: ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) - Cohort B | Up to 4.5 years
  Overall Survival (OS) defined as time from first dose of 1st line treatment to death from any cause.
Overall Survival (OS) - Cohort C | Up to 4.5 years
  Overall Survival (OS) defined as time from first dose of 1st line treatment to death from any cause.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort A | At Screening - Up to 28 days after signed consent]
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort B | At Screening - Up to 28 days after signed consent]
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort C | At Screening - Up to 28 days after signed consent]
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort A | At Day 1 of Each Treatment Cycle (2-6-week cycles, per specific agent)
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort B | At Day 1 of Each Treatment Cycle (2-6-week cycles, per specific agent)
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L - Cohort C | At Day 1 of Each Treatment Cycle (2-6-week cycles, per specific agent)
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.

CONTACTS AND LOCATIONS:
Overall Officials: Liza Villaruz, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No